CLINICAL TRIAL: NCT05951036
Title: Effects of Additional Blood Flow Restriction and Sham Blood Flow Restriction in Eccentric Exercise on Muscle Strength, Dynamic Stability, and Reduce the Risk of ACL Injury
Brief Title: Effect of Blood Flow Restriction Training to Muscle Strength, Dynamic Stability, and ACL Injury Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, I Putu Gde Surya Adhitya, Principal Investigator, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1575/UN14.2.2.VII.14/LT/2023
Record Dates: First submitted 2023-07-02; First posted 2023-07-18 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects; Sports Level 1
Keywords: blood flow restriction training; sham blood flow restriction training; BFR; Eccentric training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LL-BFRt (Experimental): 30% of repetition maximum and 70% of arterial occlusion pressure
  Interventions: Procedure: Low-load Blood Flow Restriction training
- Sham LL-BFRt (Sham Comparator): 30% of repetition maximum and 10% of arterial occlusion pressure
  Interventions: Procedure: Sham Low-load Blood Flow Restriction training
- HL-Et (Active Comparator): 70% of repetition maximum
  Interventions: Procedure: High-load Eccentric training

INTERVENTIONS:
Procedure: Low-load Blood Flow Restriction training — Physical therapist will apply the BFR cuffs with 70% of arterial occlusion pressure on the both legs of participants. Then, participants will be asked to perform eccentric trainings (including, double leg squats, split squats, deadlifts, and monster walks) with 30% of repetition maximum.
  Arms: LL-BFRt
Procedure: Sham Low-load Blood Flow Restriction training — Physical therapist will apply the BFR cuffs with 10% of arterial occlusion pressure on the both legs of participants. Then, participants will be asked to perform eccentric trainings (including, double leg squats, split squats, deadlifts, and monster walks) with 30% of repetition maximum.
  Arms: Sham LL-BFRt
Procedure: High-load Eccentric training — Physical therapist will ask participants to perform eccentric trainings (including, double leg squats, split squats, deadlifts, and monster walks) with 70% of repetition maximum.
  Arms: HL-Et

SUMMARY:
The goal of this randomized clinical trial study is to compare low-load blood flow restriction (LL-BFRt), sham LL-BFRt, and high-load eccentric training (HL-Et) in healthy level 1 sportsman. The main questions it aims to answer are:

1. Does LL-BFR improve muscle strength better than sham LL-BFRt and HL-Et?
2. Does LL-BFR improve dynamic stability better than sham LL-BFRt and HL-Et?
3. Does LL-BFR prevent ACL injury better than sham LL-BFRt and HL-Et?

Participants will be randomized into three intervention groups: LL-BFRt, sham LL-BFRt, and HL-Et. Participants will be asked to do:

* In LL-BFRt, participants will be asked to do LL eccentric training (including double leg squats, split squats, deadlifts, and monster walks) with a 30% of repetition maximum (RM) and 70% of arterial occlusion pressure (AOP).
* In sham LL-BFRt, participants will be asked to do LL eccentric training with a 30% of repetition maximum (RM) and 10% of arterial occlusion pressure (AOP).
* In HL-Et, participants will be asked to do LL eccentric training with a 70% of repetition maximum (RM).

Researchers will compare LL-BFRt, sham LL-BFRt, and HL-Et to see if muscle strength, dynamic stability, and ACL injury prevention improve after the interventions and follow-up.

DETAILED DESCRIPTION:
Participants will be asked to do five sets of ten repetitions of each eccentric training, one-minute rest interval for each eccentric training and two mins rest interval between each set.

ELIGIBILITY:
Inclusion Criteria:

* Being 15-35 years old
* Perform sports level 1 (soccer, basket ball, futsal, combat martial art) at least twice per week.
* Never had an history of ACL injury
* Never had an history of sprain or strain grade III
* Agree to participate until the end of this study period and sign the inform consent

Exclusion Criteria:

* Having hypertension, blood circulation disease, anemia, obesity, diabetes, kidney failure, vena thromboembolic, cancer, and tumor.
* Disabilities or disabled people.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 8 weeks
  Investigators will measure the quadriceps muscle isometric strength using dynamometer (units: Newton or kilogram).
Dynamic stability I | 8 weeks
  Investigators will measure the dynamic stability I using Y-balance test (units: centimeter).
Dynamic stability II | 8 weeks
  Investigators will measure the dynamic stability II using single leg hop test (units: centimeter).

CONTACTS AND LOCATIONS:
Locations (1):
- Physical therapy laboratory, College of Medicine, Universitas Udayana and ROM Physiotherapy Private Clinic Denpasar, Denpasar, Bali, Indonesia

REFERENCES:
- [Derived] Adhitya IPGS, Aryana IGNW, Kurniawati I, Thanaya SAP, Utama MBR. Effect of Low-Load Blood Flow Restriction Training and High-Load Resistance Training on Quadriceps Strength, Dynamic Stability, and Functional Performance. Clin J Sport Med. 2025 Feb 11. doi: 10.1097/JSM.0000000000001330. Online ahead of print. PMID 39932234